CLINICAL TRIAL: NCT02896907
Title: A Pilot Study of Intravenous Ascorbic Acid and Folfirinox in the Treatment of Advanced Pancreatic Cancer
Brief Title: Ascorbic Acid and Combination Chemotherapy in Treating Patients With Locally Advanced or Recurrent Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.347; JT 8223 (Other: JeffTrial Number)
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; dehydroftorafur; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (FOLFIRINOX, ascorbic acid) (Experimental): Patients receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours on day 1. Patients then receive ascorbic acid IV over 2 hours on days 3, 5, 8, 10 and 12. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Fluorouracil; Dietary Supplement: Ascorbic Acid

INTERVENTIONS:
Drug: Oxaliplatin — Given IV
  Other Names: Diaminocyclohexane Oxalatoplatinum; Eloxatin; Dacotin; Dacplat; 61825-94-3; [(1R,-2R)-1,2-cyclohexanediamine-N,N'][oxalato (2--)-O,O']platinum; [Sp-4-2-(1R-trans)]-(1,2,cyclohexanediamine-N,N')[ethanedioato(2--)-O,O']platinum; Ai Heng; Oxalatoplatin; trans-l diaminocyclohexane oxalatoplatinum
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: 136572-09-3; Campto; Camptosar; Camptothecin 11
Drug: Leucovorin Calcium — Given IV
  Other Names: 1492-18-8; 3590; 5-Formyl Tetrahydrofolate; 5-Formyl-5,6,7,8-tetrahydrofolic Acid; 5-Formyl-5,6,7,8-tetrahydropteroyl-L-glutamic Acid; Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium N-(p-((((6RS)-2-amino-5-formyl-5,6,7,8-tetrahydro-4-hydroxy-6-pteridinyl)methyl)amino)benzoyl)-L-glutamate (1:1); Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Flynoken A; Folaren; Folaxin; Foliben; Folinic Acid Calcium Salt Pentahydrate; Folix; Lederfolin; Leucosar; N-[4-[[(2-Amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amnio]benzoyl]-L-glutamic Acid; Rescufolin; Tonofolin; Rescuvolin; Wellcovorin
Drug: Fluorouracil — Given IV
  Other Names: 19893; 2,4-Dioxo-5-fluoropyrimidine; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; AccuSite; Fluracedyl; Fluracil; Fluroblastin; Ribofluor; Ro 2-9757
Dietary Supplement: Ascorbic Acid — Given IV
  Other Names: 2-(1,2-dihydroxyethyl)-4,5-dihydroxy-furan-3-one; 33832; 50-81-7; Asorbicap; C Vitamin; C-Long; Ce-Vi-Sol; Cecon; Cenolate; L-Ascorbic Acid; Vitamin C

SUMMARY:
This pilot clinical trial studies the side effects of ascorbic acid and combination chemotherapy in treating patients with pancreatic cancer that has spread to other places in the body, has come back, or cannot be removed by surgery. Nutrients found in food and dietary supplements, such as ascorbic acid, may improve the tolerability of chemotherapy regimens. Drugs used in chemotherapy, such as fluorouracil, irinotecan hydrochloride, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ascorbic acid and combination chemotherapy may work better in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine safety of intravenous ascorbic acid in combination with fluorouracil, irinotecan hydrochloride, leucovorin calcium, and oxaliplatin (FOLFIRINOX) as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 in patients with advanced pancreatic cancer.

SECONDARY OBJECTIVES:

I. To test feasibility of collecting quality of life (QOL), patient reported outcomes (PRO) data and correlative studies on patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Histological diagnosis of adenocarcinoma of the pancreas
* Stage IV or recurrent pancreatic cancer by imaging
* Locally advanced unresectable pancreatic cancer by National Comprehensive Cancer Network (NCCN) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* No prior treatment for metastatic disease (prior neo-adjuvant or adjuvant chemotherapy, except FOLFIRINOX, chemoradiation or radiation allowed)
* White blood count >= 3000
* Platelets >= 100,000
* Total bilirubin =< 1.5 mg/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5 X upper limit of normal (ULN)
* Creatinine < 1.5 mg/dL
* Glucose-6-phosphatase deficiency (G6PD) level of 5-14 units/g hemoglobin (Hgb) or within institutional standard parameters
* All subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study

Exclusion Criteria:

* Other pancreatic cancer histology (islet cell, acinar, neuroendocrine tumors)
* Resectable pancreatic cancer
* Prior neoadjuvant FOLFIRINOX
* Pregnant or lactating females
* No clinical ascites (mild ascites on scans permissible)
* Central nervous system (CNS) metastasis
* Known congestive heart failure, significant ventricular arrhythmias, cirrhosis, grade 4/5 chronic kidney disease, uncontrolled diabetes
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Peripheral neuropathy grade 2 or greater
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Posey, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (FOLFIRINOX, Ascorbic Acid)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (FOLFIRINOX, Ascorbic Acid)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as Determined by CTCAE Version 4.03
Description: After 4 patients are enrolled on the study and receive at least one dose of intravenous ascorbic acid, the data will be reviewed. If 2 out of the 4 cannot complete 2 courses of FOLFIRINOX then the study will be halted.
Time Frame: Up to 28 days after the last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FOLFIRINOX, Ascorbic Acid)
Number analyzed (Participants) | 8
Participants
  Grade 4 adverse event | 1
  Grade 5 adverse event | 1
  Grade 3 adverse event | 4
  No Serious Adverse Events | 2

2. Secondary Outcome: Change in Quality of Life as Defined by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30
Description: Change in quality of life over the six measurement times will be modeled using mixed effects linear regression to account for correlation among repeated measurements from the same subjects. Average change in QoL from baseline to follow-up will be computed.
Time Frame: Baseline to up to 28 days after the last treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (FOLFIRINOX, Ascorbic Acid)
Number analyzed (Participants) | 8
score on a scale | NA (NA) — Due to the small number of participants, quality of life assessments were not looked at quantitatively. Attempts have been made to obtain additional information from the investigator but no information has been provided.

ADVERSE EVENTS:
Time Frame: baseline through 30 days after completing treatment; an average of 4 months.
Arm/Group | Treatment (FOLFIRINOX, Ascorbic Acid)
All-Cause Mortality (participants affected / at risk) | 6/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (FOLFIRINOX, Ascorbic Acid) (N=8)
Sepsis (Blood and lymphatic system disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypokalemia (General disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02896907/Prot_SAP_000.pdf